CLINICAL TRIAL: NCT03791229
Title: The Evaluation of Pain and Discomfort After Appendectomy in Children and Their Effects on Quality of Life
Brief Title: Pain and Discomfort After Appendectomy in Children
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Onur Palabiyik, Assistant Professor, Medical Doctor, Sakarya University
Other Study IDs: SAU14113
Record Dates: First submitted 2018-12-21; First posted 2019-01-02 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Appendicitis; Chronic Post-Procedural Pain
Keywords: Appendectomy; Chronic abdominal pain; Discomfort; Numerical rating scale; Pediatric quality of life inventory
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Appendectomy is the most common surgical procedure. Chronic abdominal pain is an uncommon complication following appendectomy. It is observed that pediatric patients who have undergone abdominal surgical procedure complained of pain and discomfort in the postoperative period and these complaints may affect quality of life. We aimed to investigate the presence of postoperative chronic abdominal pain and discomfort in children aged 8-18 years underwent appendectomy and their social and physical effects. The records of children aged 8-18 years who underwent appendectomy, such as age, gender, American Society of Anesthesiology (ASA) classification score, the type of surgical procedure, and anesthetic technique were obtained. Children had inclusions crietrias, pain was assessed using numerical rating scale and their effects on life were assessed Pediatric Quality of Life Inventory parent and child versions questionnaire at sixth months after surgery.

DETAILED DESCRIPTION:
Acute appendicitis is a diagnosis with clinical findings, laboratory tests and radiological imaging. The main pathology of appendicitis is usually the onset of the inflammatory process in the appendix vermiformis in the right lower abdomen. If untreated, the inflammatory process may progress to the perforation of the appendix and develop peritonitis. Appendectomy is an emergency surgical procedure for treatments of patients diagnosed with acute appendicitis and is the most common surgical procedure (1). Complications of appendectomy are wound site infection, postoperative intestinal adhesions and obstruction, peritonitis, bleeding, inguinal hernia, and chronic abdominal pain.

It is observed that pediatric patients who have undergone abdominal surgical procedure complained of pain and discomfort in the postoperative period (2). It should be noted that these complaints may affect quality of life. To the best of our knowledge, since there is no study in the literature, we aimed to investigate the presence of postoperative chronic abdominal pain and discomfort in children aged 8-18 years underwent appendectomy and their social and physical effects.

After Local Ethics Committee approval had been obtained, the records of children aged 8-18 years who underwent appendectomy, such as age, gender, American Society of Anesthesiology (ASA) classification score, the type of surgical procedure, and anesthetic technique were obtained from hospital information management system and anesthetic charts. Inclusion criterias were children between the ages of 8-18 years who underwent appendectomy, had ASA I physical score, and those who agree to participate for this research. Children who aged under 8 and over 18 years, had ASA II and those with higher physical score, had previously undergone surgery from the right lower abdomen, had preoperative pain complaint over 6 month, had psychiatric disorders, and whose parents do not agree to participate were excluded in this study. By calling parents, at the 6th month after the surgical procedure, the presence of chronic pain and discomfort were asked via face to face or talking on the phone. The primary endpoint of this study is to investigate the prevalence of chronic pain and discomfort at the 6th month after appendectomy in pediatric patients. The secondary endpoint is to determine the effects of chronic pain on the children's quality of life.

Pain was defined as the presence of intermittent or continuous hurtfully sensation. Discomfort was defined as an abnormal bad feeling. Children were asked whether they felt pain or discomfort while resting, coughing, and exercise. Pain was assessed using verbal numeric rating scale. Their effects on life were assessed Pediatric Quality of Life Inventory parent and child versions questionnaire at sixth months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 8-18 years who underwent appendectomy,
* who had ASA I physical score
* who agree to participate for this research

Exclusion Criteria:

* Children who aged under 8 and over 18 years,
* who had ASA II and those with higher physical score,
* who had previously undergone surgery from the right lower abdomen,
* who had preoperative pain complaint over 6 month,
* who had psychiatric disorders,
* who do not agree to participate

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 8-18 years who underwent appendectomy
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of chronic pain | at the 6th month after appendectomy in pediatric patients
  The primary endpoint of this study is to investigate the prevalence of chronic pain and discomfort. Chronic pain is going to be assessed using numeric rating scale (NRS). The NRS for pain is a unidimensional measure of pain intensity in adults and children. The pain NRS is a single 11-point numeric scale. An 11-point numeric scale (NRS 11) with 0 representing one pain extreme (e.g., "nopain") and 10 representing the other pain extreme (e.g.,"pain as bad as you can imagine" and "worst pain imag-inable"). 0 point represents "no pain", 1-3 "mild pain", 4-6 "moderate pain", 7-10 "severe pain".

SECONDARY OUTCOMES:
the effects of chronic pain on quality of life | at the 6th month after appendectomy in pediatric patients
  The secondary endpoint is to determine the effects of chronic pain on the children's quality of life. Pediatric Quality of Life Inventory Parent and Child Versions (PedQL-P and C) is going to apply to children which report chronic pain and discomfort for evaluating their effects on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Onur Palabiyik, MD, Principal Investigator — Sakarya University School of Medicine, Department of Anesthesiology
Locations (1):
- Sakarya University School of Medicine Department of Anesthesiology, Sakarya, Adapazari, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No